CLINICAL TRIAL: NCT01907399
Title: Study of Immune Response in Obesity and Type 2 Diabetes
Acronym: IMMUNOBEDIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Bonnotte PHRC IR 2010
Record Dates: First submitted 2013-07-17; First posted 2013-07-25 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Obesity; Type 2 Diabetes; Healthy Volunteers
Keywords: obese patients; obese patients with type 2 diabetes; healthy volunteers
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Blood Specimen Collection

ARMS (3):
- obese patients (Other): (BMI> 30 kg/m2) androids (waist circumference> 102 cm in men and> 88 cm in woman)
  Interventions: Other: Blood samples
- obese patients with type 2 diabetes (Other): (BMI> 30 kg/m2) androids (waist circumference> 102 cm in men and> 88 cm in woman)with diabetes
  Interventions: Other: Blood samples
- healthy volunteers (Other): free of disease inflammatory or infectious and will have a BMI <25 Kg/m2et fasting glucose <1g / L
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples

SUMMARY:
There is a link between activation of the immune response inducing chronic inflammation and both obesity and type 2 diabetes. To date, however, the cause(s) of this inflammation, the mechanisms of the inflammatory cascade and the type of cells involved are not completely known. The aim of our project is to study the principal cell types involved in the immune response from a quantitative and functional point of view in obese diabetic patients versus obese non-diabetic patients and healthy subjects who are neither diabetic nor obese.

Despite possible inter-individual heterogeneity of immune cells, the fact that this work will be carried out by an accredited team with considerable expertise in the study of almost all the different types of immune cells will probably make it possible to know whether cell dysfunction and inflammation are associated with obesity or rather linked to insulin resistance. This study will be completed later by a second study on cell infiltration in adipose tissues in the 3 groups defined above. Better understanding of the physiopathology and especially the mechanisms and type of cells involved in obesity-related inflammation could quickly lead to the development of appropriate therapies that could act specifically on the cells involved and thus preclude the onset of complications.

ELIGIBILITY:
Inclusion Criteria:

* Patient-control who have given written informed consent Patient-control who are covered by the National Health Insurance Agency Patient-control > 18 years old

The criteria to classify patients into groups will be as follows:

Group 1- Obese diabetics BMI > 30 Kg /m2 AND fasting glycemia > 1.26 g/L AND Triglycerides >1.5g/L AND HDL <0.4g/L (men), <0.5g/L (women) Group 2- Obese non-diabetics without metabolic syndrome BMI > 30 Kg /m2 AND fasting glycemia < 1.10 g/L AND Triglycerides <1.5g/L AND HDL >0.4g/L (men), >0.5g/L (women) Group 3- Healthy Subjects BMI < 25 Kg/m² AND fasting glycemia < 1.10g/L AND Triglycerides <1.5g/L

Exclusion Criteria:

* Persons not covered by the National Health Insurance Agency Patients who presented a recent infection, or cancer or patients treated with corticosteroids or anti-inflammatory drugs. Patients with diabetes following an overload disease (hemochromatosis) or due to a disease of the pancreas Chronic infection Pregnant women Patients on the following treatments (glitazone: Actos, Avendia; GLP1 Agonist: Byetta, Victoza; Fibrates) Patients presenting severe renal insufficiency with clearance<30ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
quantification of Treg | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France